CLINICAL TRIAL: NCT05307055
Title: Theta Burst Subthalamic Nucleus Deep Brain Stimulation for Cognitive and Motor Improvements in Parkinson's Disease
Brief Title: Evaluation of Neurocognitive Changes in Parkinson's Disease After Low Frequency Burst Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Darrin J Lee, MD, PhD, Assistant Professor of Neurological Surgery, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HS-20-00676
Record Dates: First submitted 2022-03-14; First posted 2022-04-01 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease
Keywords: Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A (Experimental): double-blinded randomization into theta burst stimulation followed by baseline stimulation
  Interventions: Device: STN DBS - Theta Burst; Device: STN DBS - Gamma
- Group B (Experimental): double blinded randomization into baseline stimulation followed by theta burst stimulation
  Interventions: Device: STN DBS - Theta Burst; Device: STN DBS - Gamma

INTERVENTIONS:
Device: STN DBS - Theta Burst — 200 Hz intraburst stimulation for 0.1 second repeated at intervals of 5hz with an existing device
Device: STN DBS - Gamma — Standard of care gamma stimulation with an existing device

SUMMARY:
This study aims to determine whether direct brain stimulation of specific regions and ranges improves cognition in people with Parkinsons Disease (PD) who already have a deep brain stimulator implanted. Research activities consist of 32 subjects undergoing stimulation changes to their device and being administered neurocognitive tests to evaluate the changes. An fMRI scan will also be done at baseline and at weeks 15 and 27.

All subjects will undergo the stimulation changes in a randomized double blind crossover study. Evaluation of stimulation changes will be assessed through analysis of neurocognitive data.

DETAILED DESCRIPTION:
In this single-center pilot study, the investigators will study both acute and chronic changes to neurocognitive and motor performance in response to interleaving gamma/theta (theta burst) stimulation compared to standard-of-care gamma stimulation.

This study will be a randomized double-blinded crossover study. Each patient's baseline voltage intensity will be unchanged. During the first outpatient visit, a baseline assessment (under baseline stimulation parameters, including frequency, pulse width and voltage) consisting of motor and cognitive tests will first be performed. After one week of titration on the theta burst stimulation paradigm, all patients will randomized to either baseline or theta burst stimulation settings for one week. Motor testing (UPDRS) and neuropsychological testing will be performed after this week. Each patient will then be programmed to the other stimulation paradigm for another week. At the end of this third week, neuropsychological and motor testing will again be performed.

Patients will again be randomized into either baseline gamma stimulation or theta burst stimulation for the chronic phase of the study. Repeat neuropsychological and motor testing will be performed at three months. Each patient will switched to the other stimulation strategy and repeat neuropsychological and motor testing will be performed after another three months. After the first 6 months, patients will be placed on open-label theta burst stimulation for 6 months (total of one year). At the end of one year, patients will undergo repeat neuropsychological and motor testing, after which they will be reprogrammed to their initial settings or given the option to remain on theta burst stimulation parameters. Functional magnetic resonance imaging will be acquired during baseline, week 15, and week 27 visits for patients with compatible devices that meet the inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients who had previously undergone bilateral STN deep brain stimulation implantation
2. Age >18 years old
3. Stable medication regimen for at least 3 months.
4. Patient informed and able to give written consent
5. Able to comply with all testing, follow-ups and study appointments and protocols

Exclusion Criteria:

1. History of epilepsy or seizure
2. History of dementia
3. History of major substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-11 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of motor symptoms | Baseline, Week 1, Week 2, Week 3, Week 15, Week 27
  Effects of theta burst stimulation on changes in baseline motor symptoms will be assessed using the MDS-Unified Parkinson's Disease Rating Scale - Sections III&IV (MDS-UPDRS III&IV)
Evaluation of executive functioning | Baseline, Week 1, Week 2, Week 3, Week 15, Week 27
  Effects of theta burst stimulation on changes in baseline cognitive symptoms will be assessed using Delis-Kaplan Executive Function System (D-KEFS).
Neuroimaging | Baseline, Week 15, Week 27
  Effects of theta burst stimulation on changes in baseline resting state functional connectivity will be assessed using functional magnetic resonance imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Darrin Lee, MD PhD, Principal Investigator — University of Southern California, Keck School of Medicine
Locations (1):
- University of Southern California Keck School of Medicine, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT05307055/ICF_000.pdf